CLINICAL TRIAL: NCT05425706
Title: Investigation of the Effectiveness of Mulligan Concept Sustained Natural Apophysial Glides (SNAGs) Technique in Non-Specific Neck Pain Patients: A Randomized Controlled Single Blinded Trial
Brief Title: Sustained Natural Apophysial Glides (SNAGs) Technique in Non-Specific Neck Pain Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Duygu Korkem, Assistant Professor, Hacettepe University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2017-KAEK-120/2019-14
Record Dates: First submitted 2022-06-08; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Neck Pain
Keywords: manual therapy; neck pain; SNAGs; sleep quality; quality of life
MeSH Terms: conditions — Neck Pain; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experiment group (Experimental): Number of participant is 16. In addition to the conventional therapy, SNAGs technique was applied.
  Interventions: Other: application of SNAGs technique
- control group (No Intervention): Number of participant is 16. Only the conventional therapy was applied.

INTERVENTIONS:
Other: application of SNAGs technique — in experiment group, the SNAGs technique was applied to 16 participants in addition to conventional therapy.
  Arms: experiment group

SUMMARY:
Mechanical neck pain is defined for the absence of cervical spinal pathologies.With the SNAGs mobile mobilization method, it reveals effective results in cases of limitation and pain in the cervical joints.Although there are studies with the Mulligan concept in the literature, studies examining the effects of the SNAGs technique on non-specific neck pain are limited.

The aim of this study is to investigate the effectiveness of the Mulligan Concept SNAGs mobilization method applied in addition to the conventional physiotherapy program in individuals with nonspecific neck pain.

DETAILED DESCRIPTION:
This study was conducted to investigate the effectiveness of Mulligan concept cervical sustained natural apophysial glides (SNAGs) mobilization method in addition to the conventional treatment program in patients with nonspecific neck pain. The study included 40 patients (18-50 years of age) with non-specific neck pain, radicular compression and loss of strength for at least 3 months, diagnosed by a specialist physician; patients with central nervous system disease, distal-peripheral nerve injuries Patients with inflammatory joint disease, cervical spine fracture or surgery, patients with upper extremity surgery, cervical spine tumor and infection, cervical spine congenital anomaly and diabetes were not included in the study. 15 sessions were applied for 3 weeks, 5 days a week for 10 weeks, 10 minutes ultrasound, 20 minutes transcutaneous electrical nerve stimulation (TENS) and hotpack application and Mulligan mobilization in addition to physiotherapy programs. The patient was rested for 5 seconds between sets. The physiotherapy program was applied to the control group and the application session was completed. Normal range of motion exercises were performed in both groups and given as home exercise.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer patients with non-specific neck pain lasting at least 3 months,
* Volunteer patients without radicular pressure,
* Volunteer patients with loss of strength,
* Volunteer patients diagnosed with non-specific neck pain by a specialist physician.

Exclusion Criteria:

* Volunteer patients with central nervous system disease,
* Volunteer patients with distal-peripheral nerve injuries,
* Volunteer patients with inflammatory joint disease,
* Volunteer patients with cervical spine fracture or surgery, upper extremity surgery,
* Volunteer patients with vertebrobasilar artery stenosis,
* Volunteer patients with osteoporosis,
* Volunteer patients with cervical dislocation,
* Volunteer patients with cervical spine tumor and infection,
* Volunteer patients with congenital anomalies involving the spine,
* Volunteer patients with patients with diabetes.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2020-01-06 (Actual); Study Completion 2020-04-06 (Actual)

PRIMARY OUTCOMES:
Range of motion assessments | Two weeks for each participants
  Active and passive range of motion
Pain assessments | Two weeks for each participants
  McGill Pain Scale; minimum pain score: 0, maximum pain score: 78, The higher the pain score the greater the pain.

SECONDARY OUTCOMES:
Sleep quality assessments | Two weeks for each participants
  Pittsburgh Sleep Quality Index (PSQI)
Quality of life assessments | Two weeks for each participants
  The Nottingham Health Profile

CONTACTS AND LOCATIONS:
Overall Officials: DUYGU KORKEM YORULMAZ, PhD., Principal Investigator — ISTINYE UNİVERSITY
Locations (1):
- Istınye University Medical Park Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ali A, Shakil-Ur-Rehman S, Sibtain F. The efficacy of Sustained Natural Apophyseal Glides with and without Isometric Exercise Training in Non-specific Neck Pain. Pak J Med Sci. 2014 Jul;30(4):872-4. PMID 25097535
- [Result] Shin EJ, Lee BH. The effect of sustained natural apophyseal glides on headache, duration and cervical function in women with cervicogenic headache. J Exerc Rehabil. 2014 Apr 30;10(2):131-5. doi: 10.12965/jer.140098. eCollection 2014 Apr. PMID 24877050